CLINICAL TRIAL: NCT02195882
Title: Effect of an Exercise Program of the Scapular Muscle Stabilizers in Amateur Kayakers Shoulder Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CEU San Pablo University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CEU-008
Record Dates: First submitted 2014-07-18; First posted 2014-07-21 (Estimated); Last update posted 2015-07-07 (Estimated); Status verified 2014-07

CONDITIONS: Shoulder Pain
Keywords: strength training; scapular stabilization; kayakers.
MeSH Terms: conditions — Shoulder Pain

ARMS (1):
- Exercise program (Experimental)
  Interventions: Procedure: Exercise program of the scapular muscle stabilizers

INTERVENTIONS:
Procedure: Exercise program of the scapular muscle stabilizers

SUMMARY:
The purpose of this study is to determine whether a specific strengthening program for the stabilizing scapular muscle can reduce shoulder pain of amateur kayaker.

ELIGIBILITY:
Inclusion Criteria:

* There Have Been practicing kayaking over 3 years.
* There Have Been shoulder pain during sports at least 1 month of evolution

Exclusion Criteria:

* Shoulder pain was caused by a traumatic injury.
* To be in medical, pharmacological or shoulder physiotherapy treatment during the study.
* To have been surgically intervened in the shoulder

Ages: 14 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 11 (Actual)
Dates: Start 2014-05; Primary Completion 2014-09 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Change in pain level during kayakergometer test | participants will be followed for the duration of kayakergometer test, an expected average of 30 minutes

SECONDARY OUTCOMES:
change in the time of appearance of the symptoms during kayakergometer test. | participants will be followed for the duration of kayakergometer test, an expected average of 30 minutes

CONTACTS AND LOCATIONS:
Locations (1):
- San Pablo CEU University, Boadilla del Monte, Madrid, Spain